CLINICAL TRIAL: NCT03837704
Title: A Controlled, Open-label, 3-arm Parallel Group, Multi-center Study to Evaluate the Abdominal Aortic Aneurysm (AAA) Growth Rate in Adult Smoking Patients Randomized to Either Cigarette Smoking or IQOS Use and to Compare With the AAA Growth Rate in Patients Who Had Stopped Smoking
Brief Title: Comparison of Abdominal Aortic Aneurysm Growth in Adult Smoking Patients Who Either Switch to IQOS, Continue Smoking, or Quit Smoking.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: P1-AAA-02-JP
Record Dates: First submitted 2019-01-21; First posted 2019-02-12 (Actual); Results first posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Smoking; Abdominal Aortic Aneurysm; IQOS Use
MeSH Terms: conditions — Smoking; Aortic Aneurysm, Abdominal | interventions — Tobacco Products

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IQOS Arm (Active Comparator): Patients diagnosed with AAA, switching from cigarette smoking to IQOS use
  Interventions: Other: IQOS
- CC Arm (Active Comparator): Patients diagnosed with AAA, continuing to smoke cigarettes
  Interventions: Other: Cigarette
- Smoking Cessation Arm (Active Comparator): Patients diagnosed with AAA, who have completely stopped smoking and are not using any other tobacco or nicotine-containing product(s)
  Interventions: Other: Smoking Cessation

INTERVENTIONS:
Other: IQOS — AAA patients will switch from cigarette smoking to ad libitum IQOS use, with no flavor variant restrictions.
  Arms: IQOS Arm
Other: Cigarette — AAA patients will continue to smoke their cigarettes ad libitum, with no brand restrictions.
  Arms: CC Arm
Other: Smoking Cessation — AAA patients who have completely quit smoking will continue to remain abstinent from smoking cigarettes or using any tobacco or nicotine-containing product(s)
  Arms: Smoking Cessation Arm

SUMMARY:
The purpose of this study was to evaluate the reduction of the Abdominal Aortic Aneurysm (AAA) annual growth rate in patients who switched from smoking cigarettes to using IQOS as compared to patients who continued to smoke cigarettes, and to patients who had quit smoking. The study also aimed to provide context to the scale of reduction in the growth rate, by comparing the AAA annual growth rates for continuing to smoke and switching to IQOS with the AAA annual growth rate in smokers who had stopped smoking. The study further evaluated the effects of switching to IQOS on co-morbidities observed in AAA patients that are related to smoking as well as to assess the effects on relevant Biomarkers of Potential Harm (BoPH) linked to smoking related diseases.

DETAILED DESCRIPTION:
This was a controlled, open-label, 3-arm parallel group, multi-center study in patients diagnosed with Abdominal Aortic Aneurysm (AAA) to evaluate the AAA annual growth rate in adult smokers randomized to either continue smoking combustible cigarettes (CC) or to switch to IQOS and in adults who had stopped smoking, as a non-randomized control arm.

This was a descriptive study, designed to gain an understanding of how changes in smoking behaviors impact AAA growth rate and disease progression. Therefore, there were no formal statistical hypotheses to be tested.

Smoking patients with AAA who did not quit smoking after their AAA diagnosis, and who were not intending to quit within the next 6 months were screened for enrollment and randomization in the CC and IQOS arms if all other eligibility criteria were met.

Smoking patients with AAA who had completely stopped smoking and using any other tobacco or nicotine-containing products within 2 months of their AAA diagnosis, and were still abstinent at the time of the Screening Visit and of the Baseline Visit were screened to be enrolled in the smoking cessation (SC) arm without randomization.

ELIGIBILITY:
General Inclusion Criteria:

* Patient diagnosed with AAA (infrarenal, fusiform type) with a current aortic maximum minor-axis diameter of 30 to ≤ 49 mm (in male patient) and 30 to ≤ 44 mm (in female patient).
* Patient has smoked on a daily basis (no brand restrictions) for at least 5 years prior to AAA diagnosis, based on self-reporting
* Patient is ready to comply with the study protocol (e.g., to use their assigned product/regimen during the course of the study)

Inclusion criteria specific to patients screened for enrollment and randomization to the CC or IQOS arm:

* Patient has smoked on average at least 5 commercially available CC per day (no brand restriction) for the last 12 months, based on self-reporting. Intermittent attempts to quit smoking not exceeding 2 months or short-term interruption of smoking up to 10 days within the last 12 months will be allowed. Smoking status will be verified based on a urinary cotinine test (i.e., cotinine ≥ 200 ng/mL).
* Not intending to quit smoking within the next 6 months after having been advised to quit smoking.

Inclusion Criteria specific to patients screened for enrollment into the SC arm:

* Patient had completely quit smoking and stopped the use of any other tobacco or nicotine-containing products within 6 months after AAA diagnosis, and is still abstinent at Screening and at Baseline. Smoking status will be verified based on a urinary cotinine test (i.e., cotinine < 100 ng/mL).

Exclusion Criteria:

* Patient is legally incompetent, physically or mentally incapable of giving consent.
* Patient is a current or former employee of the tobacco industry or their first-degree relatives (parent and child); patient is an employee of the investigational site or any other parties involved in the study or their first-degree relatives (parent and child).
* Patient has been previously screened or enrolled in this study or was enrolled in any clinical study within 3 months prior to the Screening Visit.
* Female patient who is pregnant or breast-feeding.
* Patient is ineligible as judged by the Investigator to participate in the study for any reason.
* Patient with acute severe cardiovascular events or respiratory diseases, within the last 3 months; with currently active cancer or history of cancer within the last 5 years; with dissecting aneurysm(s) of the aorta; with infrarenal pseudo-AAA (false AAA); with a diagnosis of COPD Stage 3 and 4 in the medical history; with a recent (within 1 year) or current history of alcohol or other substance abuse based on self-reporting.
* Patient with a diagnosis of concomitant genetic diseases such as but not limited to Marfan syndrome, Loeys-Dietz syndrome, Vascular Ehlers-Danlos syndrome, Turner syndrome, Polycystic kidney disease, Noonan syndrome, Alagile syndrome, Arterial tortuosity syndrome and Cutis laxa.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Jaumont, MD, Study Chair — Philip Morris Products SA
Locations (13):
- Japan (13):
  - Chiba-Nishi General Hospital, Matsudo, Chiba
  - Tokyo Bay Urayasu Ichikawa Medical Center, Urayasu, Chiba
  - Fujita General Hospital, Fujita, Fukushima
  - Kitakanto Cardiology Hospital, Shizukawa, Gunma
  - Shonan Kamakura General Hospital, Okamoto, Kamakura
  - Atsugi City Hospital, Atsugi, Kanagawa
  - AOI Universal Hospital, Kawasaki, Kanagawa
  - Shin-Yurigaoka General Hospital, Kawasaki, Kanagawa
  - Saitama Cardiovascular and Respiratory Center, Itai, Kumagaya
  - Kishiwada Tokushukai Hospital, Kishiwada, Osaka
  - Kasukabe Chuo General Hospital, Kasukabe, Saitama
  - Okitama Public General Hospital, Nanyō, Yamagata
  - Omichikai Morinomiya Hospital, Osaka

RESULTS

PARTICIPANT FLOW:
Period: Completed V3 (Month 6)
Arm/Group | IQOS Arm | CC Arm | Smoking Cessation Arm
Started | 16 | 16 | 16
Completed | 16 | 16 | 16
Not Completed | 0 | 0 | 0
Period: Completed V4 (Month 12)
Arm/Group | IQOS Arm | CC Arm | Smoking Cessation Arm
Started | 16 | 16 | 16
Completed | 16 | 16 | 15
Not Completed | 0 | 0 | 1
Period: Completed V5 (Month 18)
Arm/Group | IQOS Arm | CC Arm | Smoking Cessation Arm
Started | 16 | 16 | 15
Completed | 16 | 14 | 14
Not Completed | 0 | 2 | 1
Period: Completed V6 (Month 24)
Arm/Group | IQOS Arm | CC Arm | Smoking Cessation Arm
Started | 16 | 14 | 14
Completed | 14 | 13 | 14
Not Completed | 2 | 1 | 0
Period: Completed V7 (Month 30)
Arm/Group | IQOS Arm | CC Arm | Smoking Cessation Arm
Started | 14 | 13 | 14
Completed | 14 | 12 | 14
Not Completed | 0 | 1 | 0
Period: Completed V8 (Month 36)
Arm/Group | IQOS Arm | CC Arm | Smoking Cessation Arm
Started | 14 | 12 | 14
Completed | 13 | 11 | 14
Not Completed | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IQOS Arm | CC Arm | Smoking Cessation Arm | Total
Number analyzed (Participants) | 16 | 16 | 16 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.0 (6.19) | 70.4 (7.73) | 71.3 (2.59) | 70.9 (5.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 16 | 16 | 16 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 16 | 16 | 16 | 48
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Nationality [Count of Participants; unit: Participants]
  Japanese | 16 | 16 | 16 | 48
  Other | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: AAA Annual Growth Rate Over Time
Description: AAA annual growth rate will be measured in AAA patients who switch from smoking cigarettes to using IQOS, and AAA patients who continue to smoke CC, as compared to AAA patients who had stopped smoking. Maximum minor-axis AAA diameter in mm will be measured. Annual growth rate will be calculated by annualizing the slope of the linear regression over the available diameter measurements.
Time Frame: At 6-month intervals from baseline to V8 (month 36)
Population: Full Analysis Set (FAS) population
Measure: Mean (95% Confidence Interval); unit: (mm/year)
Arm/Group | IQOS Arm | CC Arm | Smoking Cessation Arm
Number analyzed (Participants) | 15 | 16 | 15
(mm/year) | 1.80 [0.94 to 2.66] | 1.87 [1.33 to 2.40] | 1.27 [0.84 to 1.70]

2. Secondary Outcome: Percentage of Subjects Without Open Surgical AAA Treatment or AAA Endovascular Repair Over Time
Description: This outcome measured the percentage of subjects without surgery or endovascular repair over time in AAA patients who switch from smoking CC to using IQOS, as compared to AAA patients who continue smoking CC and AAA patients who had stopped smoking.
Time Frame: From time of AAA diagnosis (prior to study participation) until V8 (month 36), a time frame of up to 7 years
Population: Full Analysis Set (FAS) population
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | IQOS Arm | CC Arm | Smoking Cessation Arm
Number analyzed (Participants) | 15 | 16 | 16
percentage
  Baseline -36 months | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]
  Baseline -24 months | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 87.5 [58.6 to 96.7]
  Baseline -12 months | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 87.5 [58.6 to 96.7]
  V2 (Baseline) | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 87.5 [58.6 to 96.7]
  V4 (Month 12) | 83.9 [49.4 to 95.7] | 80.0 [40.9 to 94.6] | 87.5 [58.6 to 96.7]
  V6 (Month 24) | 83.9 [49.4 to 95.7] | 80.0 [40.9 to 94.6] | 87.5 [58.6 to 96.7]
  V8 (Month 36) | 83.9 [49.4 to 95.7] | 80.0 [40.9 to 94.6] | 87.5 [58.6 to 96.7]

3. Secondary Outcome: Percentage of Subjects Without Open Surgical AAA Treatment or AAA Rupture Over Time
Description: This outcome measured the percentage of subjects without surgery or AAA rupture over time in AAA patients who switch from smoking CC to using IQOS, as compared to AAA patients who continue smoking CC and AAA patients who had stopped smoking.
Time Frame: From time of AAA diagnosis (prior to study participation) until V8 (month 36), a time frame of up to 7 years
Population: Full Analysis Set (FAS) population
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | IQOS Arm | CC Arm | Smoking Cessation Arm
Number analyzed (Participants) | 15 | 16 | 16
percentage
  Baseline -36 months | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]
  Baseline -24 months | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]
  Baseline -12 months | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]
  V2 (Baseline) | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]
  V4 (Month 12) | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]
  V6 (Month 24) | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]
  V8 (Month 36) | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]

4. Secondary Outcome: Incidence of Open Surgical AAA Treatment or AAA Endovascular Repair and AAA Rupture
Description: The incidence of open surgical AAA treatment or AAA endovascular repair and AAA rupture will be measured in AAA patients who switch from smoking CC to using IQOS, as compared to AAA patients who continue to smoke CC and AAA patients who had stopped smoking. Incidence rate will be calculated annually.
Time Frame: From baseline to V8 (month 36)
Population: Full Analysis Set (FAS) population
Measure: Number; unit: events per person-year
Arm/Group | IQOS Arm | CC Arm | Smoking Cessation Arm
Number analyzed (Participants) | 15 | 16 | 16
events per person-year
  Number of patients with open surgical AAA treatment or endovascular repair annually | 0.05 | 0.05 | 0.05
  Number of patients with AAA rupture annually | 0.00 | 0.00 | 0.00

5. Secondary Outcome: Incidence of AAA Growth Above 5 mm Within 6 Months
Description: Incidence of AAA growth above 5 mm within 6 months will be measured in AAA patients who switch from smoking CC to using IQOS, as compared to AAA patients who continue smoking CC and AAA patients who had stopped smoking. Incidence rate will be calculated annually by counting the number of patients with an increase in maximum minor-axis AAA diameter of more than 5 mm within 6 months.
Time Frame: At 6-month intervals from baseline to V8 (month 36)
Population: Full Analysis Set (FAS) population
Measure: Number (95% Confidence Interval); unit: events per person-year
Arm/Group | IQOS Arm | CC Arm | Smoking Cessation Arm
Number analyzed (Participants) | 15 | 16 | 16
events per person-year | 0 [0.0 to 0.2] | 0 [0.0 to 0.2] | 0 [0.0 to 0.2]

6. Secondary Outcome: AAA Patients With an Overall Maximum Minor-axis AAA Diameter of >55mm in Male Patients and >50mm in Female Patients
Description: The number of AAA patients with an overall maximum minor-axis AAA diameter >55mm in male AAA patients and >50mm in female AAA patients will be counted in AAA patients who switch from smoking CC to using IQOS, as compared to AAA patients who continue smoking CC and AAA patients who had stopped smoking. (Note that the 95% CI is calculated by exact method (Clopper-Pearson) and refers to CI for a proportion).
Time Frame: From baseline to V8 (month 36)
Population: Full Analysis Set (FAS) population
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | IQOS Arm | CC Arm | Smoking Cessation Arm
Number analyzed (Participants) | 15 | 16 | 16
participants | 0 [0.0 to 0.2] | 0 [0.0 to 0.2] | 0 [0.0 to 0.2]

7. Secondary Outcome: Systolic Blood Pressure
Description: This cardiovascular BoPH (systolic blood pressure) will be measured in AAA patients who switch from smoking CC to using IQOS, AAA patients who continue to smoke CC and AAA patients who had stopped smoking.
Time Frame: From V1 (screening) to V8 (month 36)
Population: Full Analysis Set (FAS) population
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | IQOS Arm | CC Arm | Smoking Cessation Arm
Number analyzed (Participants) | 16 | 16 | 16
mmHg
  V1 (Screening) | 134.8 [126.6 to 143.0] | 128.0 [119.1 to 136.9] | 124.0 [117.1 to 130.9]
  V2 (Baseline) | 132.5 [122.9 to 142.1] | 128.9 [120.1 to 137.8] | 135.9 [129.7 to 142.2]
  V3 (Month 6) | 138.8 [129.0 to 148.6] | 131.1 [123.8 to 138.5] | 130.3 [121.5 to 139.0]
  V4 (Month 12) | 132.7 [125.5 to 140.0] | 135.0 [128.5 to 141.5] | 129.3 [121.2 to 137.5]
  V5 (Month 18) | 133.9 [125.9 to 141.9] | 130.6 [124.6 to 136.7] | 126.9 [120.0 to 133.9]
  V6 (Month 24) | 136.6 [127.3 to 146.0] | 129.7 [120.7 to 138.7] | 128.1 [121.1 to 135.2]
  V7 (Month 30) | 128.8 [121.1 to 136.5] | 136.1 [130.5 to 141.7] | 126.0 [114.1 to 137.9]
  V8 (Month 36) | 131.7 [124.6 to 138.8] | 131.6 [126.2 to 137.1] | 125.3 [116.5 to 134.0]

8. Secondary Outcome: Urinary Nicotine Equivalents (NEQ)
Description: To measure nicotine exposure over time in AAA patients who switch from smoking CC to using IQOS, AAA patients who continue to smoke CC, and AAA patients who had stopped smoking. (NEQ adjusted for creatinine (mg/g creat)).
Time Frame: From baseline to V8 (month 36)
Population: Full Analysis Set (FAS) population. Some participants were excluded from analysis for protocol deviations (including, but not limited to, missing measurements).
Measure: Geometric Mean (95% Confidence Interval); unit: mg/g creat
Groups:
- Smoking Cessation Arm: Patients diagnosed with AAA, who have completely stopped smoking and are not using any other tobacco or nicotine-containing product(s) Smoking Cessation: AAA patients who have completely quit smoking will continue to remain abstinent from smoking cigarettes or using any tobacco or nicotine-containing product(s)
Arm/Group | IQOS Arm | CC Arm | Smoking Cessation Arm
Number analyzed (Participants) | 15 | 16 | 16
mg/g creat
  V2 (Baseline) | 5.70 [4.22 to 7.72] | 6.30 [4.16 to 9.54] | 0 [0 to 0]
  V3 (Month 6) | 5.13 [4.06 to 6.47] | 7.46 [5.39 to 10.32] | 0 [0 to 0]
  V4 (Month 12): number analyzed (Participants) | 15 | 16 | 15
  V4 (Month 12) | 4.30 [2.43 to 7.61] | 5.50 [3.16 to 9.59] | 0 [0 to 0]
  V5 (Month 18): number analyzed (Participants) | 15 | 16 | 14
  V5 (Month 18) | 5.86 [3.18 to 10.78] | 0.0 [0.0 to 0.0] | 0 [0 to 0]
  V6 (Month 24): number analyzed (Participants) | 15 | 16 | 14
  V6 (Month 24) | 4.65 [2.70 to 8.02] | 4.32 [1.97 to 9.48] | 0 [0 to 0]
  V7 (Month 30): number analyzed (Participants) | 15 | 16 | 14
  V7 (Month 30) | 3.88 [2.22 to 6.78] | 4.24 [1.98 to 9.07] | 0 [0 to 0]
  V8 (Month 36): number analyzed (Participants) | 15 | 16 | 14
  V8 (Month 36) | 0 [0 to 0] | 4.20 [1.46 to 12.07] | 0 [0 to 0]

9. Secondary Outcome: Diastolic Blood Pressure
Description: This cardiovascular BoPH (diastolic blood pressure) will be measured in AAA patients who switch from smoking CC to using IQOS, AAA patients who continue to smoke CC and AAA patients who had stopped smoking.
Time Frame: From V1 (screening) to V8 (month 36)
Population: Full Analysis Set (FAS) population.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | IQOS Arm | CC Arm | Smoking Cessation Arm
Number analyzed (Participants) | 16 | 16 | 16
mmHg
  V1 (Screening) | 75.4 [69.6 to 81.1] | 76.6 [71.0 to 82.2] | 72.9 [67.5 to 78.4]
  V2 (Baseline) | 76.6 [70.5 to 82.6] | 76.6 [71.5 to 81.6] | 77.3 [73.0 to 81.5]
  V3 (Month 6) | 79.7 [75.0 to 84.3] | 77.3 [73.4 to 81.2] | 73.9 [68.1 to 79.6]
  V4 (Month 12) | 76.3 [70.5 to 82.2] | 77.3 [70.8 to 83.7] | 74.1 [68.0 to 80.1]
  V5 (Month 18) | 74.8 [69.2 to 80.4] | 78.3 [72.4 to 84.2] | 71.5 [67.4 to 75.6]
  V6 (Month 24) | 79.0 [74.3 to 83.7] | 78.5 [71.6 to 85.5] | 72.7 [68.3 to 77.1]
  V7 (Month 30) | 76.3 [72.5 to 80.1] | 79.8 [73.9 to 85.6] | 69.2 [62.9 to 75.5]
  V8 (Month 36) | 73.8 [68.0 to 79.5] | 77.8 [70.7 to 84.9] | 67.0 [61.5 to 72.5]

10. Secondary Outcome: Body Weight
Description: This cardiovascular BoPH (body weight) will be measured in AAA patients who switch from smoking CC to using IQOS, AAA patients who continue to smoke CC and AAA patients who had stopped smoking.
Time Frame: From V1 (screening) to V8 (month 36)
Population: Full Analysis Set (FAS) population
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | IQOS Arm | CC Arm | Smoking Cessation Arm
Number analyzed (Participants) | 16 | 16 | 16
kg
  V1 (Screening) | 68.44 [61.68 to 75.19] | 66.63 [60.48 to 72.78] | 67.91 [62.34 to 73.48]
  V2 (Baseline) | 68.13 [61.51 to 74.75] | 66.61 [60.47 to 72.74] | 67.93 [62.39 to 73.47]
  V3 (Month 6) | 67.79 [61.04 to 74.54] | 65.88 [60.00 to 71.76] | 67.98 [62.56 to 73.40]
  V4 (Month 12) | 68.47 [61.53 to 75.42] | 66.51 [60.42 to 72.59] | 67.27 [61.38 to 73.16]
  V5 (Month 18) | 69.41 [62.02 to 76.81] | 67.60 [61.22 to 73.98] | 66.70 [60.47 to 72.93]
  V6 (Month 24) | 68.51 [62.41 to 74.61] | 67.82 [60.19 to 75.45] | 67.14 [61.06 to 73.21]
  V7 (Month 30) | 67.61 [61.70 to 73.53] | 69.08 [61.79 to 76.38] | 66.03 [59.84 to 72.22]
  V8 (Month 36) | 68.74 [62.36 to 75.12] | 69.71 [61.56 to 77.86] | 66.34 [59.61 to 73.08]

11. Secondary Outcome: Waist Circumference
Description: This cardiovascular BoPH (waist circumference) will be measured in AAA patients who switch from smoking CC to using IQOS, AAA patients who continue to smoke CC and AAA patients who had stopped smoking.
Time Frame: From V1 (screening) to V8 (month 36)
Population: Full Analysis Set (FAS) population
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | IQOS Arm | CC Arm | Smoking Cessation Arm
Number analyzed (Participants) | 16 | 16 | 16
cm
  V1 (Screening) | 90.51 [85.59 to 95.44] | 90.30 [85.11 to 95.49] | 91.40 [86.57 to 96.23]
  V2 (Baseline) | 89.88 [84.61 to 95.14] | 91.01 [85.10 to 96.91] | 93.33 [88.80 to 97.85]
  V3 (Month 6) | 89.95 [84.90 to 95.00] | 89.91 [84.06 to 95.75] | 91.16 [86.50 to 95.81]
  V4 (Month 12) | 89.75 [84.17 to 95.34] | 89.46 [84.39 to 94.54] | 91.78 [86.74 to 96.82]
  V5 (Month 18) | 91.73 [86.60 to 96.85] | 90.71 [84.99 to 96.42] | 91.82 [86.81 to 96.83]
  V6 (Month 24) | 89.14 [81.91 to 96.36] | 91.55 [84.13 to 98.97] | 91.54 [86.91 to 96.16]
  V7 (Month 30) | 89.04 [84.25 to 93.82] | 93.33 [86.51 to 100.16] | 91.43 [86.59 to 96.27]
  V8 (Month 36) | 91.78 [87.65 to 95.90] | 92.30 [85.63 to 98.97] | 91.36 [85.93 to 96.79]

12. Secondary Outcome: Total 4-(Methylnitrosamino)-1-(3-pyridyl)-1-butanol (Total NNAL)
Description: This biomarker of exposure to a tobacco smoke constituent will be measured in AAA patients who switch from smoking CC to using IQOS, AAA patients who continue to smoke CC and AAA patients who had stopped smoking.
Time Frame: From baseline to V8 (month 36)
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mg creat
Arm/Group | IQOS Arm | CC Arm | Smoking Cessation Arm
Number analyzed (Participants) | 15 | 16 | 16
pg/mg creat
  V2 (Baseline): number analyzed (Participants) | 15 | 15 | 16
  V2 (Baseline) | 124.09 [81.11 to 189.85] | 87.34 [55.98 to 136.27] | 0 [0 to 0]
  V3 (Month 6): number analyzed (Participants) | 14 | 16 | 16
  V3 (Month 6) | 39.83 [17.74 to 89.41] | 108.70 [73.72 to 160.27] | 0 [0 to 0]
  V4 (Month 12): number analyzed (Participants) | 13 | 16 | 15
  V4 (Month 12) | 27.12 [10.69 to 68.83] | 81.24 [52.33 to 126.12] | 0 [0 to 0]
  V5 (Month 18): number analyzed (Participants) | 14 | 14 | 14
  V5 (Month 18) | 32.81 [12.77 to 84.33] | 61.85 [33.78 to 113.27] | 0 [0 to 0]
  V6 (Month 24): number analyzed (Participants) | 13 | 13 | 14
  V6 (Month 24) | 33.02 [12.70 to 85.89] | 57.78 [31.17 to 107.11] | 0 [0 to 0]
  V7 (Month 30): number analyzed (Participants) | 13 | 12 | 14
  V7 (Month 30) | 27.54 [10.09 to 75.21] | 61.78 [31.22 to 122.26] | 0 [0 to 0]
  V8 (Month 36): number analyzed (Participants) | 12 | 10 | 14
  V8 (Month 36) | 35.24 [12.12 to 102.43] | 42.36 [15.30 to 117.29] | 0 [0 to 0]

13. Secondary Outcome: Total N-nitrosonornicotine (Total NNN)
Description: as for outcome 12
Time Frame: From baseline to V8 (month 36)
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mg creatinine
Arm/Group | IQOS Arm | CC Arm | Smoking Cessation Arm
Number analyzed (Participants) | 15 | 16 | 16
pg/mg creatinine
  V2 (Baseline): number analyzed (Participants) | 15 | 15 | 16
  V2 (Baseline) | 3.26 [1.78 to 5.97] | 2.09 [1.00 to 4.38] | 0 [0 to 0]
  V3 (Month 6): number analyzed (Participants) | 14 | 16 | 16
  V3 (Month 6) | 1.39 [0.73 to 2.68] | 2.86 [1.61 to 5.09] | 0 [0 to 0]
  V4 (Month 12): number analyzed (Participants) | 13 | 16 | 14
  V4 (Month 12) | 0.98 [0.42 to 2.30] | 2.12 [1.00 to 4.49] | 0 [0 to 0]
  V5 (Month 18): number analyzed (Participants) | 14 | 14 | 13
  V5 (Month 18) | 1.28 [0.50 to 3.28] | 1.47 [0.54 to 4.00] | 0 [0 to 0]
  V6 (Month 24): number analyzed (Participants) | 13 | 12 | 14
  V6 (Month 24) | 1.34 [0.51 to 3.52] | 1.55 [0.51 to 4.68] | 0 [0 to 0]
  V7 (Month 30): number analyzed (Participants) | 13 | 12 | 14
  V7 (Month 30) | 1.20 [0.44 to 3.24] | 1.31 [0.50 to 3.48] | 0 [0 to 0]
  V8 (Month 36): number analyzed (Participants) | 12 | 10 | 14
  V8 (Month 36) | 1.10 [0.37 to 3.27] | 1.27 [0.37 to 4.41] | 0 [0 to 0]

14. Secondary Outcome: 2-cyanoethylmercapturic Acid (2-CyEMA)
Description: as for outcome 12
Time Frame: From baseline to V8 (month 36)
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mg creat
Arm/Group | IQOS Arm | CC Arm | Smoking Cessation Arm
Number analyzed (Participants) | 15 | 16 | 16
ng/mg creat
  V2 (Baseline): number analyzed (Participants) | 15 | 15 | 16
  V2 (Baseline) | 95.38 [71.93 to 126.48] | 98.95 [64.68 to 151.37] | 2.36 [1.36 to 4.10]
  V3 (Month 6): number analyzed (Participants) | 13 | 16 | 16
  V3 (Month 6) | 20.21 [8.29 to 49.27] | 111.31 [74.30 to 166.76] | 1.67 [0.99 to 2.81]
  V4 (Month 12): number analyzed (Participants) | 13 | 16 | 15
  V4 (Month 12) | 13.29 [4.61 to 38.34] | 82.46 [51.19 to 132.83] | 2.30 [1.10 to 4.80]
  V5 (Month 18): number analyzed (Participants) | 14 | 14 | 14
  V5 (Month 18) | 12.53 [4.58 to 34.27] | 56.77 [26.94 to 119.63] | 1.70 [0.82 to 3.51]
  V6 (Month 24) | 13.88 [4.22 to 45.68] | 48.40 [18.83 to 124.44] | 1.77 [0.77 to 4.06]
  V7 (Month 30) | 8.25 [2.72 to 24.99] | 52.08 [20.21 to 134.23] | 1.51 [0.76 to 3.01]
  V8 (Month 36) | 12.32 [3.31 to 45.91] | 46.19 [13.07 to 163.23] | 1.86 [0.92 to 3.77]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the signature of the ICF by each subject until the end of the safety follow-up period, a total duration for each subject of up to 37 months.
Arm/Group | IQOS Arm | CC Arm | Smoking Cessation Arm
All-Cause Mortality (participants affected / at risk) | 1/16 | 1/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 3/16 | 5/16 | 7/16
Other Adverse Events (participants affected / at risk) | 14/16 | 13/16 | 14/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IQOS Arm (N=16) | CC Arm (N=16) | Smoking Cessation Arm (N=16)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Inflammatory pseudotumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tarsal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IQOS Arm (N=16) | CC Arm (N=16) | Smoking Cessation Arm (N=16)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Pterygium (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Oropharyngeal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (6)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tooth loss (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis allergic (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Contrast media allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Morphoea (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Urticaria (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Dermatophytosis of nail (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes ophthalmic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1) | 3 (3)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Tinea infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (3) | 4 (9)
Viral uveitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (3)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Occult blood positive (Investigations) | 0 (0) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (2)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0)
Gastrointestinal submucosal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Progressive supranuclear palsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Chest discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Carotid artery stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness postural (Vascular disorders) | 0 (0) | 1 (3) | 0 (0)
Hypertensions (Vascular disorders) | 1 (1) | 4 (4) | 3 (3)
Varicose vein (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (4) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This was an exploratory study not powered to detect a difference in AAA diameter between the different study arms. Due to patient recruitment challenges, only 48 patients out of the 114 planned were enrolled and the study was shortened from 5 to 3 years. Due to the limited sample size potential confounders could also not be adjusted for.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
We confirm we have the contractual provisions in place which specify that in no event will the study site be allowed to disclose to any third party (or publicly release) any information obtained through the study without the CRO's prior written consent which in turn cannot provide such consent without Sponsor's approval unless such publication is made to satisfy regulatory requirements.

The Intellectual Property rights and research results from the present study belong to the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2021-09-17): https://cdn.clinicaltrials.gov/large-docs/04/NCT03837704/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-20): https://cdn.clinicaltrials.gov/large-docs/04/NCT03837704/SAP_001.pdf